CLINICAL TRIAL: NCT00410241
Title: ClinSeq: A Large-Scale Medical Sequencing Clinical Research Pilot Study
Status: Active, not recruiting | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070002; 07-HG-0002
Record Dates: First submitted 2006-12-09; First posted 2006-12-12 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-09-09

CONDITIONS: Healthy Volunteers; Atherosclerotic Heart Disease
Keywords: Genome; Cardiovascular; Volunteers; Genes; Atherosclerosis; Natural History
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- A1: Self-referred individuals 45-65 at enrollment, 25% of whom had coronary artery disease
- A2: Individuals 45-65 at enrollment who self-identified as African, African-American, or Afro-Caribbean
- A3: Adults aged 18-65 at the time of enrollment, including subjects of both sexes, who have been identified as likely to return for follow up
- B: Family members of Group A1, A2, or A3

SUMMARY:
This study will examine genome sequencing in clinical research. Genome sequencing is a process in which researchers analyze (or sequence) part or all of the genome from a single person. The human genome is the material in cells that includes thousands of genes. Gene changes that cause or contribute to disease can be passed on from one generation to the next. This study first focuses on heart disease. Later, researchers hope to study other conditions and genes, with the eventual goal of sequencing most or all of participants genes.

Participants ages 45 to 65 years of age and who do not smoke, may be eligible for this study. Patients will come to the NIH Clinical Research Center for an initial study to last about half a day. They will donate a blood sample and complete a short survey. Then they will meet the genetic counselor to learn more about genome sequencing. Those who join the study will undergo the following procedures and evaluations:

* Family history and medical history.
* Measurement of height and blood pressure.
* Noninvasive heart tests, including electrocardiogram and echocardiogram.
* Drawing of about 3 ounces of blood (5 to 6 tablespoons); part of the blood sample will be used for research and another part for clinical testing.
* Multidetector computed tomography (CT), a test to measure coronary artery calcification, that is, condition of inflexibility.

Each patient will receive a letter with results of the clinical laboratory values and evaluations. There will be recommendations for follow-up with the patient s doctors. Risks in this study include exposure to radiation from the CT test. The radiation amount used is about the same that a person normally receives from natural sources, such as from the sun, outer space, and radioactive materials found naturally in the earth s air and soil. Another slight risk involves reactions to a contrast agent that may be used in the echocardiogram. Side effects can be headache, nausea or vomiting, a warm sensation, and dizziness.

With the samples that patients provide, researchers will start by sequencing about 400 genes related to heart disease. Analysis will take months to complete. Genome sequencing is difficult to do, and researchers have much to learn about the genes they sequence and the gene changes they find. If the researchers find gene changes that are important to the health of a participant, they will contact that participant and give him/her the choice of learning such results.

This study may or may not have a direct benefit for participants. Patients would get free clinical testing for cholesterol, diabetes, and other conditions, as well as information about gene changes. Knowledge gained will benefit people in the future as researchers learn about the relationship between gene changes and health.

DETAILED DESCRIPTION:
The purpose of ClinSeq is to research large-scale medical sequencing (LSMS) in a clinical research setting. It was developed at a time (approximately 2007) when little was known about the processes and outcomes of doing so. By conducting LSMS and returning individual results to participants, we intended to investigate some of the technical, medical, and genetic counseling issues that accompanied the implementation of LSMS in the clinical setting. Three of our objectives have been met and the relevant findings have largely been published including:

* Developing methods for recruiting and consenting a large, racially-diverse cohort
* Continuing to improve upon existing algorithms for generating and interpreting sequence data
* Build and offer this cohort as a resource for addressing biomedical research questions including investigating the association of genomic variants with traits and phenotypes

However, there is still much to be learned regarding LSMS, much of which is pertinent to our original aim of improving our understanding of socio-behavioral aspects of implementation of LSMS in a clinical research setting. Remaining objectives include:

* To understand patient outcomes (e.g., health behavior, communication, personal utility, emotional) following the receipt of medically actionable results.
* To investigate the impact of an intervention designed to promote better understanding of the

accuracy of genetic sequencing among those consenting to LSMS.

* To investigate the outcomes of returning negative secondary findings reports via a website and compare two versions of a slide developed to improve women s understanding of their residual risk for breast cancer following the receipt of such a report.
* To identify genetic risk factors for diabetes and other metabolic diseases related to glucose metabolism.

ELIGIBILITY:
* INCLUSION CRITERIA:

Group A

Recruitment and enrollment to Group A is complete. For the most part, the same inclusion and exclusion criteria and justifications applied to the A1, A2, and A3 cohorts, but exceptions have been noted for some criteria. Overall, those criteria included:

-Criterion #1 (A1): 25% of the participants in this cohort have known coronary artery disease (CAD), which is defined as history of: myocardial infarction, silent myocardial infarction, stent placement, re-vascularization, 50% or more arterial blockage, a calcium

score greater than the 95th centile based on their age, gender and race (using the MESA calculator at www.mesa-nhlbi.org/Calcium), or a strong family history of CAD along with a personal history of a potentially CAD-related biochemical phenotype, such as elevated

lipoprotein (a) (Lp(a)).

* Justification: Because CAD was initially the target phenotype under study, it was critical to include a minimal number of participants with documented disease.

  * Criterion #2 (A1 & A2): Individuals eligible for this study are required to be non-smokers at the time of enrollment, for our purposes defined as someone who has not smoked regularly during the previous 12 months (Wilson et al., 1998).
* Justification: Because our study originally aimed to identify the genetic underpinnings of CAD, we excluded individuals who were smokers because it is a significant, known risk factor for CAD.

  -Criterion #3 (A1 and A2): Individuals without CAD must be 45-65 years of age, and individuals with CAD must be 35-65 years of age.
* Justification: We selected our age range based on the manifestations of our target phenotype. We selected the lower limit of this cutoff in order to recruit a cohort whose coronary artery calcification (CAC) measurements range from normal to diseased, and it has been shown that abnormal CAC is infrequent below this age (Janowitz, Agatston, Kaplan, & Viamonte, 1993). The lower limit of the age range

has been expanded in the case of CAD participants to allow for the enrollment of individuals with particularly severe personal or family history of cardiovascular disease. An upper age limit of 65 was chosen to allow for longitudinal study of participants.

-Criterion #4 (A3): Individuals must be 18-65 years of age.

* Justification: As with the A1 and A2 cohort, an upper age limit of 65 was chosen to allow for longitudinal study of participants. However, in contrast to the A1 and A2 cohorts, a lower age limit of 18 was chosen because we are no longer primarily interested in a cardiovascular disease phenotype.

  -Criterion #5 (All Cohorts): Subjects must reside in the metropolitan DC and Baltimore areas or travel to the CRC on a regular basis for follow-up, or be willing to travel to the NIH as needed for protocol participation at their own expense (with the exception of some participants with CAD who had extremely compelling personal or family history of disease and we agreed to cover the cost of their transportation, meals and lodging covered for clinical visits because they could not otherwise participate).
* Justification: This criterion is designed to minimize subjects reluctance to participate in ongoing study activities, such as ancillary studies and return to receive genetic testing results.

  -Criterion #6: First-degree relatives of enrolled ClinSeq participants are not eligible unless they fall into Group B.
* Justification: These individuals share on average 50% of their genes on autosomal loci, thus possibly reducing the power of a study, such as ClinSeq , with a focus on common diseases.

  * Criterion #7: Individuals who are directly involved with gathering and analyzing the clinical and genotyping data, including the Principal Investigator, the Associate Investigators, the ClinSeq staff involved with the subjects at the clinical level (such as the Nurse Practitioner, Genetic counselor, etc.), and the staff at NISC involved with generating and analyzing the sequence data are ineligible.
* Justification: Participation of these individuals may present a conflict of interest (COI) and lead to adverse events (AEs).

  -Criterion #9: Individuals who are already enrolled in another study that provides genome or exome sequencing, such as the GENE-FORECAST Study (14-HG_0048) are ineligible.
* Justification: The results that we provide will no longer be needed by the participant. In addition, the results will no longer be novel to the participant, making them ineligible for all social and behavioral research aimed at understanding the impact of return of results. Because this severely limits their participation in the project, we propose to exclude these participants.

  -Criterion #11: Adults who cannot or may become unable to consent are excluded from this study.
* Justification: Because the study is interested in learning how people make consent decisions, their attitudes, and use of personal testing results, these individuals are excluded from the project.

The following participants are/were eligible for projects related to Objectives 1A-C & 2:

* Objective 1A: Participants eligible for this project must be over 18 years old and have received a medically actionable genetic result in the last six months.

  --Justification: Only individuals with a result can be interviewed and surveyed because we are interested in their experiences.
* Objective 1B: Recruitment and data collection are complete. Eligibility criteria included: (1) consenting to the ClinSeq project between 2012-2018, (2) completion of the Baseline Survey, and (3) being over 18 years old.
* Objective 1C: Recruitment and data collection are complete. Eligibility for inclusion in this project were based on: (1) having a negative secondary finding report available from exome sequence data analysis, and (2) consenting to participate in a randomized control trial of results return.

  * Justification: Only participants with negative secondary findings results were included in the study since the project is focused initially on return of these results only.

Objective 2: Recruitment and data collection are complete. Participants eligible for this group had a variant of interest identified in a gene/genes related to diabetes or other metabolic diseases related to glucose metabolism.

--Justification: We are interested in understanding whether specific genetic variants have phenotypic consequences thus, having a variant is required for inclusion of a subject s data in our dataset.

Group B

Recruitment and enrollment to Group B is closed. The eligibility for Group B was distinct from Group A. Group B eligibility required:

-Criterion #1: Having a relative enrolled in Group A

--Justification: There are were two justifications for including relatives in Group B of the study. The first is that we wished to initiate standard of care approaches for known disease entities. For example, it is clinically indicated to perform family studies of relatives of persons with familial hypercholesterolemia to identify persons at high risk for this life-threatening disorder. The second was that we may

sometimes needed additional genetic data on the families to help us determine if a genetic variant is associated with a disease phenotype (both in cases where we had some evidence of the link between the variant and disease thus the variant was suspected to cause disease and in cases where we had little to no evidence of such a link thus the variant may cause disease).

-Criterion #2: Being over 18 years old, unless the phenotype under study affects children

--Justification: We excluded children unless the disease causes symptoms in childhood because of our concern that such genetic testing could pose a risk to these children without known benefit.

EXCLUSION CRITERIA:

No Exclusion as the recruitment and enrollment is closed.

Ages: 6 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants in Groups A reside in the local area or were willing to return up to once per year at their own expense and be the age of 45-65 (or 18-65 for A3) unless they have a significant personal/family history of coronary artery disease, in which case we also accepted individuals age 35-65. Participants in Group B were invited to the study by the team and were family members of Group A1, A2, or A3 participants.
Sampling Method: Non-Probability Sample
Enrollment: 1665 (Actual)
Dates: Start 2007-01-05 (Actual)

PRIMARY OUTCOMES:
Recruit & consent cohort | 2017
  Developing methods for recruiting and consenting a large, racially-diverse cohort
Offer cohort as resource | 2026
  Build and offer this cohort as a resource for addressing biomedical research questions including investigating the association of genomic variants with traits and phenotypes
Improvement to algorithms for interpreting sequence data | 2026
  Continuing to improve upon existing algorithms for generating and interpreting sequence data
Health behavior, family communication and understanding | 2026
  Determining the impacts of LSMS results on health behaviors, family communication and understanding
Efficiency of result disclosure | 2026
  Piloting increasingly efficient models for returning LSMS results

CONTACTS AND LOCATIONS:
Overall Officials: Leslie G Biesecker, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (2):
- United States (2):
  - Suburban Hospital, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: Yes
We are actively depositing data into the database of genotypes and phenotypes (dbGaP), which is designed with tiered access to clinical data. That is, there is open, public access to summary clinical data of study participants and qualified investigators may apply for access to individual, coded clinical results. Such access is limited to authorized med researchers and redistribution and security policies are strict. Broad future use of the data deposited into dbGaP (as opposed to restricted use for specific disorders) will be permitted.@@@@@@Sequence traces for individual genes will be available publicly (deposited in GenBank); however, these sequence traces won't be linked to a participant's identifiable information, nor to the sequence traces of other genes sequenced in that participant's sample.@@@@@@Coded genomic data are available to data contributors and NIH intramural investigators through the Reverse Phenotyping Core browser (18-HG-0129; https://tgac.nhgri.nih.gov/).
Supporting Information: Study Protocol
Time Frame: Data in dbGap is stored per NIH policy. Data in the Reverse Phenotyping Core/TGAC browser will be stored for the remainder of the protocol (18-HG-0129) and the time the study is closed, a proposal to the IRB will be made to keep the data or destroy it.
Access Criteria: dbGap is a controlled-access database with view-only access to summary-level information and individual-level genotype and sequence data associated with phenotypic features. The Reverse Phenotyping Core/TGAC browser allows researchers to identify particular genotypes or ranges of genotypes, while preserving the privacy of study participants by only displaying aggregate data for one or a limited number of loci in a search. The browser is located on NIH servers and searchable only by investigators in the NIH s intramural research program or external collaborators who have contributed sequence data.

REFERENCES:
- [Background] Panganamala RV, Sharma HM, Sprecher H, Geer JC, Cornwell DG. A suggested role for hydrogen peroxide in the biosynthesis of prostaglandins. Prostaglandins. 1974 Oct 10;8(1):3-11. doi: 10.1016/0090-6980(74)90031-8. No abstract available. PMID 4457956
- [Background] Freed ED, Miller A. An analysis of a continuing medical education questionnaire sent to psychiatrists in the Southern Transvaal. S Afr Med J. 1979 Aug 4;56(5):177-80. PMID 45060
- [Background] Huggenvik JI, Craven CM, Idzerda RL, Bernstein S, Kaplan J, McKnight GS. A splicing defect in the mouse transferrin gene leads to congenital atransferrinemia. Blood. 1989 Jul;74(1):482-6. PMID 2752125
- [Derived] Chan PA, Lewis KL, Biesecker BB, Erby LH, Fasaye GA, Epps S, Biesecker LG, Turbitt E. Preferences for and acceptability of receiving pharmacogenomic results by mail: A focus group study with a primarily African-American cohort. J Genet Couns. 2021 Dec;30(6):1582-1590. doi: 10.1002/jgc4.1424. Epub 2021 Apr 19. PMID 33876469
- [Derived] Biesecker BB, Lewis KL, Umstead KL, Johnston JJ, Turbitt E, Fishler KP, Patton JH, Miller IM, Heidlebaugh AR, Biesecker LG. Web Platform vs In-Person Genetic Counselor for Return of Carrier Results From Exome Sequencing: A Randomized Clinical Trial. JAMA Intern Med. 2018 Mar 1;178(3):338-346. doi: 10.1001/jamainternmed.2017.8049. PMID 29356820
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2007-HG-0002.html